CLINICAL TRIAL: NCT01754532
Title: Correlation Between Clinical Deterioration in Schizophrenic Patients and Hair Cortisol Levels
Status: Completed | Type: Observational
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Aviv Segev, Resident, Shalvata Mental Health Center
Other Study IDs: SHA-12-0028
Record Dates: First submitted 2012-12-12; First posted 2012-12-21 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Schizo-Affective Disorder
Keywords: Schizophrenia; Schizo-Affective Disorder; Stress; Cortisol; PANSS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10mg of posterior vertex hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schizophrenia patients
  Interventions: Biological: Hair Sample

INTERVENTIONS:
Biological: Hair Sample — Analysis of hair cortisol levels

SUMMARY:
The importance of stress as a possible deteriorating factor for schizophrenic patients is well documented. However, this notion is based on subjective experience and retrospective psychological analysis.

A novel method of measuring cortisol using hair has a proven correlation to subjective stress in non-clinical as well as psychiatric clinical populations.

This pilot study will attempt to assess the use of cortisol hair level, as a marker of stress, to predict clinical deterioration in schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Diagnosis of schizophrenia or schizoaffective disorder, made by a senior psychiatrist.
* Signing an informed consent.

Exclusion Criteria:

* Additional psychiatric diagnosis
* Boldness or hair shorter than 1cm
* Physiological disturbance in the HPA or the use of steroidal medication
* Neurological disease (past or present) or neurosurgery.
* Pregnancy
* Substantial chronic physical diseases/

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with Schizophrenia or Schizo-Affective Disorder
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Positive And Negative Symptoms Score | 3 month
  correlation between hair cortisol level change from baseline and PANSS score change from baseline.
Change from Baseline in Positive And Negative Symptoms Score | 6 month
  correlation between hair cortisol level change from baseline and PANSS score change from baseline.

SECONDARY OUTCOMES:
Change from Baseline in SANS, CGI, CDS, GAF and QOL Scores | 3 month
  correlation between hair cortisol level change from baseline and SANS, CDS, GAF, CGI, and QOL scores change from baseline.
Change from Baseline in SANS, CGI, CDS, GAF and QOL Scores | 6 month
  correlation between hair cortisol level change from baseline and SANS, CDS, GAF, CGI, and QOL scores change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Segev, MD, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel